CLINICAL TRIAL: NCT04280328
Title: An Open-Label Study of Ciforadenant in Combination With Daratumumab in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Ciforadenant in Combination With Daratumumab in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corvus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPI-444-003
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ciforadenant; daratumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ciforadenant in combination with daratumumab (Experimental): Ciforadenant 100 mg orally twice daily in combination with daratumumab IV 16 mg/kg.
  Interventions: Drug: Ciforadenant; Drug: daratumumab

INTERVENTIONS:
Drug: Ciforadenant — 100 mg orally twice daily for 28-day cycles
  Other Names: CPI-444
Drug: daratumumab — 16 mg/kg administered intravenously as follows based on 28-day cycles:
  * Cycles 1 - 2: Days 1, 8, 15, and 22
  * Cycles 3 - 6: Days 1 and 15
  * Cycles 7 - 24: Day 1

SUMMARY:
This is a Phase 1b open-label study of ciforadenant, an oral, small molecule inhibitor targeting adenosine-2A receptors (A2AR), on safety/tolerability and efficacy in combination with daratumumab, a monoclonal antibody targeting CD38, in relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory myeloma.
* Must have been exposed to at least 2 cycles of an IMiD containing regimen and PI containing regimen and must be refractory to at least one of the two.
* Must have completed and tolerated 2 cycles of daratumumab or other anti-CD38 targeting antibodies.
* Active myeloma requiring systemic treatment.
* Measurable disease per protocol.
* ECOG performance status of 0 - 2.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* POEMS syndrome; non-secretory myeloma (no measurable protein on sFLC assay); amyloidosis.
* History of select prior malignancies.
* Previous intolerance to daratumumab or any study drug.
* Received an allogeneic stem cell transplant within 12 months, or an autologous stem cell transplant within 6 months, or have ongoing toxicity related to transplant.
* Have an active infection or serious comorbid medical condition.
* Any live attenuated vaccination against infectious diseases (e.g., influenza, varicella) within 4 weeks of initiation of study treatment; uncontrolled human immunodeficiency virus, or positive tests for hepatitis B or hepatitis C.
* Female participants pregnant or breast-feeding.
* Screening chemistry and blood counts within protocol limits
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment or anticipation of need for systemic immunosuppressant medication during study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ciforadenant in combination with daratumumab relapsed / refractory multiple myeloma. | From start of treatment to end of treatment, up to 24 months
  Incidence of treatment-emergent adverse events, as assessed by NCI CTCAE v.5
Safety and tolerability of ciforadenant in combination with daratumumab relapsed / refractory multiple myeloma. | 28 days following first administration of ciforadnenat in combination with daratumumab
  Incidence of dose-limiting toxicities (DLTs) of CPI-444 in combination with daratumumab

SECONDARY OUTCOMES:
Overall response rate. | From start of treatment to end of treatment, up to 24 months
  According to international myeloma working group guidelines (including stringent complete response [sCR], complete response [CR], very good partial response [VGPR], partial response [PR]).
Duration of response. | From start of treatment to end of treatment, up to 24 months
  Time from the first assessment showing objective response to the date of documented disease progression.
Disease control rate. | From start of treatment to end of treatment, up to 24 months
  Proportion of participants achieving disease control for ≥ 3 months.
Time to next therapy. | Up to 2 years after end of treatment.
  Time from end of treatment to starting next anti-myeloma therapy.
Progression free survival. | Up to 2 years after end of treatment.
  Proportion of participants remaining progression free or surviving at a given time.
Minimal Residual Disease. | From start of treatment to end of treatment, up to 24 months
  Rate of molecular minimal residual disease (MRD) negativity.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Strahs, Study Director — Corvus Pharmaceuticals
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States